CLINICAL TRIAL: NCT04543942
Title: Neurobiological Factors Underlying Sex Differences in Risk for Alcohol Abuse
Brief Title: Sex Differences in Risk for Alcohol Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Fillmore (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Mark Fillmore, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 50301; K01AA024519-06 (NIH)
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Abuse
Keywords: brain activation during response inhibition; BARI; fMRI; stop signal task; sex difference; menstrual; inhibitory control
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alcohol, then saline, then alcohol, then saline (Experimental): Participants first received alcohol (60mg%) intravenously and then 24-48 hours later they received saline intravenously. Two weeks later, they again received alcohol (60mg%) intravenously and then 24 - 48 hours later they received saline intravenously.
  Interventions: Drug: Alcohol; Drug: Saline
- Saline, then alcohol, then saline, then alcohol (Experimental): Participants first received saline intravenously and then 24-48 hours later they received alcohol (60mg%) intravenously. Two weeks later, they again received saline intravenously and then 24 - 48 hours later they received alcohol (60mg%) intravenously.
  Interventions: Drug: Alcohol; Drug: Saline

INTERVENTIONS:
Drug: Alcohol — Alcohol will be administered by IV infusion (60mg%).
Drug: Saline — Saline is administered as the placebo

SUMMARY:
This study will determine the neural and hormonal mechanisms underlying sex differences in sensitivity to the disinhibiting effects of alcohol in heavy drinkers.

DETAILED DESCRIPTION:
Alcohol abuse inflicts enormous physical, emotional, and financial burdens on the individual and society at large. Knowing who is at risk for alcohol abuse, and why, is crucial for the development of effective prevention and treatment strategies. Alcohol abuse has been traditionally considered a male-oriented problem and as a consequence research on risk factors specific to women has been minimal. However, the sex gap in substance abuse is closing rapidly, and findings from both animal and human studies suggest that females are actually more vulnerable to drug use than males. As such, there is an urgent need to identify sex differences in risk factors for alcohol abuse in order to develop sex-specific prevention and treatment efforts. One clear candidate risk factor is poor inhibitory control, both in terms of baseline levels of inhibition and sensitivity to the disinhibiting effects of alcohol. Recent studies suggest that sex hormones affect inhibitory control in drug-free individuals, potentially contributing to sex differences in baseline levels of inhibition. However, the degree to which fluctuations in sex hormones influence sex differences in inhibition-related brain function in sober and intoxicated individuals is not known. The proposed project will determine the neural and hormonal mechanisms underlying sex differences in sensitivity to the disinhibiting effects of alcohol in heavy drinkers.

The overall objective of the research is to identify hormonal determinants of alcohol effects on brain activation during response inhibition (BARI) in young adult female and male drinkers. BARI will be assessed using functional magnetic resonance imaging (fMRI) during performance of the stop signal task. This task reliably activates right-lateralized prefrontal regions implicated in inhibitory control. This study will assess BARI during IV alcohol (60mg%) and saline infusion in women during the early follicular and mid-luteal phases and in men at matched intervals.

ELIGIBILITY:
Inclusion Criteria:

* heavy drinking
* Alcohol Use Disorder Identification Test score above 7
* right-handed
* BMI between 19 and 26
* high school education
* fluent in English
* women must have regular menstrual cycles
* not using hormonal contraceptives

Exclusion Criteria:

* drug use disorder (SCID, DSM-5), other than nicotine or caffeine
* meets withdrawal criteria
* history of physical or psychiatric disease
* contraindication for fMRI
* pregnant or breastfeeding
* smoking more than 5 cigarettes per day

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fillmore, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University Of Kentucky Psychology Research Lab, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (2-3 Days)
Arm/Group | Alcohol, Then Saline, Then Alcohol, Then Saline | Saline, Then Alcohol, Then Saline, Then Alcohol
Started | 13 | 15
Completed | 11 | 13
Not Completed | 2 | 2
Not completed — Scheduling conflict | 2 | 2
Period: Interval Period (2 Weeks)
Arm/Group | Alcohol, Then Saline, Then Alcohol, Then Saline | Saline, Then Alcohol, Then Saline, Then Alcohol
Started | 11 | 13
Completed | 10 | 12
Not Completed | 1 | 1
Not completed — scheduling conflict | 1 | 1
Period: Second Intervention (2-3 Days)
Arm/Group | Alcohol, Then Saline, Then Alcohol, Then Saline | Saline, Then Alcohol, Then Saline, Then Alcohol
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol, Then Saline, Then Alcohol, Then Saline | Saline, Then Alcohol, Then Saline, Then Alcohol | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.7 (1.8) | 23.1 (2.3) | 23.4 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 10 | 8 | 18
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Brain Activation During Response Inhibition (BARI) - Alcohol Infusion
Description: Brain activation during response inhibition (BARI) was assessed using blood oxygenation level dependent (BOLD) fMRI during performance of the stop signal task during alcohol (60mg%) infusion. Values were determined by the contrast of BOLD activation during successful inhibition trials relative to go trials.
Time Frame: During two alcohol sessions which could occur on two of four possible days: 1 or 2 and 15 or 16; data from the two alcohol sessions are averaged together
Measure: Mean (Standard Deviation); unit: BOLD activation
Groups:
- Males: Males who received alcohol infusion (60mg%) in either day 1 and 15 or day 2 and 16 of the study.
- Females: Females who received alcohol infusion (60mg%) on either day 1 and 15 or day 2 and 16 of the study.
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
BOLD activation | 1.83 (1.11) | 2.41 (1.35)

2. Primary Outcome: Brain Activation During Response Inhibition (BARI) - Saline Infusion
Description: Brain activation during response inhibition (BARI) was assessed using blood oxygenation level dependent (BOLD) fMRI during performance of the stop signal task during saline infusion. Values were determined by the contrast of BOLD activation during successful inhibition trials relative to go trials.
Time Frame: During two saline (placebo) sessions which could occur on two of four possible days: 1 or 2 and 15 or 16; data from the two saline sessions are averaged together
Measure: Mean (Standard Deviation); unit: BOLD activation
Groups:
- Males: Males who received saline infusion in either day 1 and 15 or day 2 and 16 of the study.
- Females: Females who received saline infusion in either day 1 and 15 or day 2 and 16 of the study.
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
BOLD activation | 1.32 (1.44) | 2.64 (1.90)

3. Secondary Outcome: Estradiol Levels - Alcohol Infusion
Description: Estradiol levels (pg/mL) were measured from blood samples following alcohol infusion.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
pg/mL | 21.5 (3.2) | 71.3 (28.8)

4. Secondary Outcome: Estradiol Levels - Saline Infusion
Description: Estradiol levels (pg/mL) were measured from blood samples following saline infusion.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
pg/mL | 23.5 (7.0) | 63.3 (34.0)

5. Secondary Outcome: Progesterone Levels - Alcohol Infusion
Description: Progesterone levels (ng/mL) were measured from blood samples prior to alcohol infusion.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
ng/mL | 0.28 (0.07) | 4.1 (1.7)

6. Secondary Outcome: Progesterone Levels - Saline Infusion
Description: Progesterone levels (ng/mL) were measured from blood samples following saline infusion.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
ng/mL | 0.29 (0.09) | 3.81 (1.95)

7. Secondary Outcome: Testosterone Levels - Alcohol Infusion
Description: Testosterone levels (ng/dL) were measured from blood samples following alcohol infusion.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
ng/dL | 544.7 (252.8) | 39.0 (22.8)

8. Secondary Outcome: Testosterone Levels - Saline Infusion
Description: Testosterone levels (ng/dL) were measured from blood samples following saline infusion.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
ng/dL | 454.61 (161.04) | 23.7 (6.73)

9. Secondary Outcome: Biphasic Alcohol Effects Score - Stimulation - Alcohol Infusion
Description: The Biphasic Alcohol Effects Scale (BAES) is a 14-point self-reporting, unipolar adjective rating scale designed to measure both stimulant and sedative effects of alcohol. Scores range from 0-10 for each of the 7 Stimulation sub-scale questions, for a total Stimulation score range of 0-70. Higher scores indicate increased stimulation. This outcome measure was collected during alcohol (60mg%) infusion.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
score on a scale | 32.2 (11.5) | 23.8 (13.3)

10. Secondary Outcome: Biphasic Alcohol Effects Score - Sedation - Alcohol Infusion
Description: The Biphasic Alcohol Effects Scale (BAES) is a 14-point self-reporting, unipolar adjective rating scale designed to measure both stimulant and sedative effects of alcohol. Scores range from 0-10 for each of the 7 Sedation sub-scale questions, for a total Sedation score range of 0-70. Higher scores indicate increased sedation. This outcome measure was collected during alcohol (60mg%) infusion.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Females: Females who received alcohol infusion (60mg%) in either day 1 and 15 or day 2 and 16 of the study.
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
score on a scale | 13.8 (4.7) | 16.3 (15.3)

11. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Stimulation - Saline Infusion
Description: The Biphasic Alcohol Effects Scale (BAES) is a 14-point self-reporting, unipolar adjective rating scale designed to measure both stimulant and sedative effects of alcohol. Scores range from 0-10 for each of the 7 Stimulation sub-scale questions, for a total Stimulation score range of 0-70. Higher scores indicate increased stimulation. This outcome measure was collected during saline infusion.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
score on a scale | 25.1 (13.1) | 16.9 (11.3)

12. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Sedation - Saline
Description: The Biphasic Alcohol Effects Scale (BAES) is a 14-point self-reporting, unipolar adjective rating scale designed to measure both stimulant and sedative effects of alcohol. Scores range from 0-10 for each of the 7 Sedation sub-scale questions, for a total Sedation score range of 0-70. Higher scores indicate increased stimulation. This outcome measure was collected during saline infusion.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
score on a scale | 7.7 (9.5) | 8.9 (10.1)

13. Secondary Outcome: Drug Effects Questionnaire Score - Feel - Alcohol Infusion
Description: The Drug Effects Questionnaire (DEQ) consists of four questions to assess acute subjective response to alcohol intake. This measure captures the amount someone feels the effects of alcohol, on a scale from 0 to 100. Higher scores indicate greater levels of 'feel alcohol'. Scores were obtained during alcohol (60mg%) infusion.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
Score on a scale | 73.4 (7.6) | 61.7 (19.5)

14. Secondary Outcome: Drug Effects Questionnaire Score - Like - Alcohol Infusion
Description: The Drug Effects Questionnaire (DEQ) consists of four questions to assess acute subjective response to alcohol intake. This measure captures the amount someone likes the effects of alcohol, on a scale from 0 to 100. Higher scores indicate greater levels of 'like alcohol'. Scores were obtained during alcohol (60mg%) infusion.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
Score on a scale | 83.4 (12.5) | 65.4 (17.0)

15. Secondary Outcome: Drug Effects Questionnaire (DEQ) - Feel - Saline Infusion
Description: The Drug Effects Questionnaire (DEQ) consists of four questions to assess acute subjective response to alcohol intake. This measure captures the amount someone feels the effects of alcohol, on a scale from 0 to 100. Higher scores indicate greater levels of 'feel alcohol'. Scores were obtained during saline infusion.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
score on a scale | 11.8 (15.3) | 8.3 (14.2)

16. Secondary Outcome: Drug Effects Questionnaire (DEQ) - Like - Saline Infusion
Description: The Drug Effects Questionnaire (DEQ) consists of four questions to assess acute subjective response to alcohol intake. This measure captures the amount someone likes the effects of alcohol, on a scale from 0 to 100. Higher scores indicate greater levels of 'like alcohol'. Scores were obtained during saline infusion.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Males | Females
Number analyzed (Participants) | 9 | 13
score on a scale | 50.5 (7.4) | 48.8 (2.9)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at each of the four study visits over approximately 4 weeks of study participation.
Groups:
- Males: Males who received alcohol or saline infusions on day 1, 2, 15, or 16 of the study.
- Females: Females who received alcohol or saline infusions on day 1, 2, 15, or 16 of the study.
Arm/Group | Males | Females
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT04543942/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT04543942/ICF_000.pdf